Official Title: A web-based intuitive eating intervention for young women with disordered eating: A pilot randomized controlled trial

**NCT number:** not yet assigned

**Date of document: 2/15/2021** 

### Introduction

Over the past 20 years, average adult weight and BMI has risen in the United States (U.S.), sparking a rise in public and private efforts to improve health via weight loss and dietary change [17, 20, 21]. Though a great deal of time and money has been dedicated to this, average BMI has not decreased and health has not improved [2, 4, 27, 29, 33]. However, the fight against weight gain has been linked to severe unintended consequences including weight cycling, distraction from health goals, increased rates of weight stigmatization, body dissatisfaction, disordered eating, and even death from extreme diets, eating disorders, weight loss surgery complications, and suicide related to these issues [2, 4, 29, 33].

Particularly, increased rates of eating disorders and disordered eating (DE) resulting from this weight-centric paradigm warrant further attention. Eating disorders carry the highest mortality rate of any mental illness, and are associated with high morbidity and societal burden [11, 12, 18, 28]. In 2019, over 10,000 people died from an eating disorder, and from 2018 to 2019 eating disorders cost the U.S. healthcare system approximately \$64.7 billion [12]. In the past 20 years, the lifetime prevalence of eating disorders in the U.S. has more-than doubled [19]. Parallel to the upsurge in eating disorders, the prevalence of DE, a subclinical pattern of maladaptive eating behavior, has also increased [30, 31]. DE is the greatest predictor for the development of an eating disorder [28]. DE disproportionately effects women, particularly young women [31, 41]. Currently, DE effects about 75% of U.S. women, most of whom will never receive treatment [7, 25, 31].

Concern for the lack of success and unintended consequences of a weight-centric paradigm has inspired calls for a shift in the promotion of healthy eating behavior. Given the high prevalence of DE, promotion of healthy eating ought to focus on this. At the forefront of this is Intuitive Eating (IE), a weight-neutral approach. The philosophy of IE posits that humans are born with the ability (an "intuition") to self-regulate appetite and make dietary choices based on internal hunger and fullness cues, but external messaging about food and body size undermines this ability and causes distress and disorder around food [35, 37]. IE is characterized by attending to internal bodily cues, and flexible thinking and behavior concerning food [35, 37]. The Intuitive Eating Scale (IES-2) provides a way to quantify IE as a construct by measuring respondents' ability to tune into various internal bodily cues [35]. In this scale, IE is broken down into 4 principles: Unconditional Permission to Eat (UPE), Reliance on Hunger and Fullness Cues (HFC), Eating for Physical Rather than Emotional Reasons (PRE), and Body-Food Choice Congruence (BFCC) [37]. Each principle is a measurable component of this style of eating; UPE is the absence of guilt or shame around eating, HFC is the ability to eat when hungry and stop when full, PRE is the ability to distinguish between physical and emotional hunger cues, and BFCC is the ability to eat in ways that are congruent with positive physical and emotional sensations and outcomes [35, 37]. These abilities are not static, though; several intervention studies have demonstrated individuals' ability to learn how to eat intuitively e.g. [7, 10, 40].

A systematic literature review of 16 IE interventions found consistent decreases in DE, depression, and increases in self-esteem [9]. While all interventions included in this review yielded improved relationship with food, mixed results were shown for weight loss, dietary changes, and physiological indicators of health [9]. Another review of 20 IE interventions demonstrated similar findings [34]. Across interventions, there were overall decreases in depression, anxiety, restriction, body dissatisfaction, and drive for thinness, and increases in self-esteem and quality of life [34]. Measures of improved physiological health including weight loss, lowered blood glucose, and lowered cholesterol levels had less data support [34].

Likewise, research examining correlates of IE reliably suggests that IE is associated with lower rates of DE, lower body preoccupation, internalized weight stigma, and rates of depression, and greater self-esteem, and quality of life [6, 7, 9, 10, 15, 34, 39, 40]. Moreover, some studies have linked IE to improved dietary quality, weight stability, and lower BMI [1, 3, 14, 16, 22, 24, 26, 32, 36, 39].

Recently, an eight-year study following 1,491 participants demonstrated strong and lasting effects of IE [15]. This study followed participants from early adolescence to young adulthood and found that both baseline levels of IE and change in IE over time predicted lower odds of depression, low self-esteem, body dissatisfaction, unhealthy weight control behaviors (fasting, skipping meals), extreme weight

control behaviors (diet pills, purging), and binge eating at follow-up [15]. The data seems to suggest that IE is a protective factor for developing DE.

Though there is strong evidence suggesting that IE is associated with lower levels of DE, few studies have examined the effect of learning to eat intuitively for people with DE. One recent study tested an uncontrolled pilot feasibility trial of a brief IE intervention for college women with DE [7]. Seventy-one women with DE participated in this first-of-its-kind intervention, demonstrating that this population can learn to eat intuitively and benefit from it [7]. Participants had medium to large improvements in IE, body appreciation, and life satisfaction, as well as reductions in DE, body dissatisfaction, and weight-bias internalization [7].

This present study is the first randomized controlled trial (RCT) testing an IE intervention for DE. This study tested various health outcomes in a web-based intervention provided to a sample of young women with DE. Participants were assessed before (time 1/T1) and after (time 2/T2) completing the intervention. T1 to T2 changes in IE, DE, body appreciation, psychological flexibility, dichotomous thinking around food, and food intake were assessed.

### **Study Aims & Hypotheses**

This study's aims were as follows: *Aim 1:* To introduce IE to a group of women with high levels of DE and assess associated outcomes. *Hypothesis 1:* When compared to the control group, the treatment group will experience the following changes from T1 to T2: (a) Increase in levels of IE, as measured by the Intuitive Eating Scale (IES-2), (b) Decrease in levels of DE, as measured by the Revised Three-Factor Eating Questionnaire (TFEQ-r18), (c) Increase in body appreciation, as measured by the Body Appreciation Scale (BAS-2), (d) Increase in psychological flexibility, as measured by the Acceptance and Action Questionnaire (AAQ-2), (e) Decrease in dichotomous thinking around food, as measured by the Dichotomous Thinking Scale (DT). *Aim 2:* To elucidate the effect of IE on food choice. *Hypothesis 2:* When compared to the control group, the treatment group's intake of fruits and vegetables, as measured by the NHANES Food Frequency Questionnaire, will increase from T1 to T2. *Hypothesis 3:* At baseline, IE will correlate with greater fruit and vegetable intake.

#### Method

### **Sample Characteristics**

Participants were women ages 18-30 from the United States and Canada with high levels of DE, defined as higher-than-average scores (score > 25) on the TFEQ-r18, without a current eating disorder diagnosis, who have never previously participated in a formal intervention or course on IE (n=123). BMI at baseline ranged from 16.3 to 65. The sample was largely college-educated, white, and heterosexual (Table 1).

Potential participants were recruited via social media and online forums, including Facebook, Instagram, Tumblr, and Reddit. Recruited participants were asked to send the study screener to others who may be interested in participating, as well. Five-hundred-thirteen completed the screener, where 390 were excluded. Some met multiple criteria for exclusion, though none were excluded for having low TFEQ-r18 scores (Figure 1).

All participant information was deidentified, and contact information was kept in a separate secured file. Each participant was assigned a unique code used to connect data from different timepoints.

At Time 1 (T1), participants were randomly assigned to either a treatment (n=62) or waitlist control group (n=61). In most aspects, the groups were not significantly different at baseline (Table 1).

### **Procedures**

IRB approval was granted from Western IRB on April 8th, 2020 (WIRB Tracking ID 20200516). After participants were recruited, the intervention began on April 29th, 2020 and concluded July 1st, 2020.

The intervention was a novel 10-week program aimed at promoting IE through pre-recorded videos, reading material, and bi-weekly discussion sessions. The intervention introduced the following

modules sequentially: Unconditional Permission to Eat, Reliance to Hunger and Fullness Cues, Body-Food Choice Congruence, Gentle Nutrition, and Joyful Movement.

Every other week, a new module was introduced. Participants were taught the concept of this module through video and reading, then prompted to practice it over the week. On opposite weeks, the module last introduced was discussed in greater detail through video, and participants were given the opportunity to discuss amongst one another and have all questions answered by the researchers. The intervention schedule included the following:

- Week 1: What is Intuitive Eating? A Program Overview and Introduction to Unconditional Permission to Eat (video + reading)
- Week 2: Discussion on Unconditional Permission to Eat, and Concerns about Eating Intuitively (video + discussion and questions/answer with researchers)
- Week 3: Reliance on Internal Cues: Eating when I'm Hungry & Stopping when I am Full (video + reading)
- Week 4: Discussion on Internal Cues, Concerns, and Questions Moving Forward -- It's OK to Make Mistakes (video + discussion and questions/answer with researchers)
- Week 5: Body-Food Choice Congruence: What Foods Make Me Feel Good? (video + reading)
- Week 6: Discussion on Food Choice -- How Do I Know if a Food Truly Makes Me Feel Good or if I Feel Good Because of Diet Culture Messages? (video + discussion and questions/answer with researchers)
- Week 7: Gentle Nutrition: Nourishing Yourself (video + reading)
- Week 8: Discussion on Nourishment, and Saying "NO" to the Food Police (video + discussion and questions/answer with researchers)
- Week 9: Joyful Movement: Find What Makes You Happy (video + reading)
- Week 10: Closing Discussion, and Final Questions (video + discussion and questions/answer with researchers)

#### Measures

## **Intuitive Eating Scale (IES-2)**

The IES-2 was administered as a pre- and post-study measure of IE skills at T1 and T2. This 21- item scale measures the extent to which a respondent follows IE principles [37]. Response options are on a 5-point Likert-type scale, with 1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree. There are four subscales on this questionnaire, each measuring a separate aspect of IE: Unconditional Permission to Eat (UPE), Reliance on Hunger and Fullness Cues (HFC), Eating for Physical Rather Than Emotional Reasons (PRE), and Body-Food Choice Congruence (BFCC). Means are calculated for overall and subscale scores. A sample item is "I trust my body to tell me when to stop eating" [37].

# National Health and Nutrition Examination Survey Food Frequency Questionnaire (N-FFQ)

The National Health and Nutrition Examination Survey Food Frequency Questionnaire (N-FFQ) was administered as a pre- and post-study measure of diet. The N-FFQ is a standardized food frequency questionnaire in which respondents are asked to recall their food and beverage intake from the past three days. It measures consumption of whole grains, refined grains, vegetables, greens, whole fruits, total fruits, total protein, plant protein, dairy, fat, sodium, added sugar, and alcohol [13].

# **Three-Factor Eating Questionnaire (TFEQ-r18)**

The TFEQ-r18 was initially used as a screening tool, then was administered post-study at T2. Higher scores on this measure indicate greater levels of pathology and distress around eating. This 18-item measure is divided into three sub-sections, each measuring a different aspect of eating distress and pathology: cognitive restraint/restriction, uncontrolled/binge eating, and emotional eating. There are six questions for cognitive restraint/restriction, nine for uncontrolled eating, and three for emotional eating. Response options are on a 4-point Likert-type scale, with 1=definitely false, 2=mostly false, 3=mostly

true, 4=definitely true. Overall and subscale scores are calculated by summing item responses. One sample item is "When I feel lonely, I console myself by eating" [23].

# **Body Appreciation Scale (BAS-2)**

The BAS-2 was used as a pre- and post-study measure of participants' body appreciation. Body appreciation is an aspect of body image that specifically targets bodily respect and contentment. The BAS-2 is a 13-item questionnaire with 5-point Likert-type scale response options, 1=never, 2=seldom, 3=sometimes, 4=often, 5=always. One sample item is "Despite its imperfections, I still like my body" [38].

#### Acceptance and Action Questionnaire (AAQ-2)

The AAQ-2 was administered as a pre- and post-study measure of psychological flexibility. The AAQ-2 directly measures behavioral effectiveness as a proxy for psychological flexibility; this is one of the most common ways to measure psychological flexibility. There are seven items, with 7-point Likert-type scale response options, 1=never true, 2=very seldom true, 3=seldom true, 4=sometimes true, 5=frequently true, 6=almost always true, 7=always true. A sample item is "I worry about not being able to control my worries and feelings" [5].

# **Dichotomous Thinking Around Food Scale (DT)**

The Dichotomous Thinking Around Food Scale (DT) was administered as a pre- and post-study measure of psychological flexibility specific to food. It is an 11-item measure of the extent to which respondents dichotomously categorize foods in an inflexible manner. Response options are on a 4-point Likert-type scale, 1=not at all true of me, 2=slightly true of me, 3=fairly true of me, and 4=very true of me. A sample item is "I think of food as either 'good' or 'bad" [8].

### **Analyses**

All analyses were completed using SPSS v.21. The data were visually inspected and cleaned prior to running analyses. Independent Sample T-Tests were used to test baseline group differences. Correlations were run for other baseline data. To test the effect of the intervention, a 2x2 analysis of variance (ANOVA) was used.

# **Data Analysis Plan**

Baseline correlations and pre- to post-study between groups analyses will be completed to test effects of IE. Correlation analyses will also be run testing associations between IE, body appreciation, psychological flexibility, dichotomous thinking around food, DE, subtypes of DE, BMI, and food choice broken down by food group. These analyses will utilize responses from all 123 participants.

At T2, 58.5% of the overall sample completed testing (n=72), including 51.6% of the treatment group (n=32), and 65.6% of the control group (n=40). Independent sample t-tests were run to compare treatment participants who completed the intervention to those who dropped out. At baseline, participants who completed treatment had higher levels of IE (t=-2.11, p=.039) and body appreciation (t=-2.39, p=.02), and lower levels of DE (t=3.5, p=.001) and dichotomous thinking (t=2.68, p=.009). There were no differences in treatment completion for participant age, race, nationality, sexual orientation, marital status, education, BMI, eating disorder history, or psychological flexibility.

To test the effect of participating in the intervention, a 2x2 ANOVA will be completed. Group x Time comparisons will examine T1 to T2 differences in the treatment and control groups.

Table 1. Participant Demographics x Group

| | Overall (n=123) | Intervention (n=62) | Control (n=61) | p |
|---|---|---|---|---|
| Median Age (years) | $25 \pm 5$ | $25 \pm 4$ | $25 \pm 6$ | .917 |
| Nationality | | | | |
| United States | 106 (86.2%) | 51 (82.3%) | 55 (90.2%) | .011* |
| Canada | 17 (13.8%) | 11 (17.7%) | 6 (9.8%) | .011* |
| Race | | | | |
| White | 86 (69.9%) | 48 (77.4%) | 38 (62.3%) | .089 |
| Asian | 10 (8.2%) | 6 (9.7%) | 4 (6.6%) | .400 |
| Latina | 7 (5.7%) | 1 (1.6%) | 6 (9.8%) | .021* |
| Black | 4 (3.3%) | 1 (1.6%) | 3 (4.9%) | .454 |
| Other | 2 (1.6%) | 0 (0%) | 2 (3.3%) | .153 |
| 2 or more races | 14 (11.3%) | 6 (9.7%) | 8 (13.1%) | .454 |
| <b>Sexual Orientation</b> | | | | |
| Heterosexual | 86 (69.9%) | 47 (75.8%) | 39 (63.9%) | .154 |
| Homosexual | 0 (0%) | 0 (0%) | 0 (0%) | 1 |
| Bisexual | 33 (26.8%) | 13 (21%) | 20 (32.8%) | .141 |
| Other | 3 (2.4%) | 2 (3.2%) | 1 (1.6%) | .572 |
| Prefer Not to Say | 1 (0.8%) | 0 (0%) | 1 (1.6%) | .315 |
| Marital Status | | | | |
| Never married | 87 (70.7%) | 43 (69.4%) | 44 (72.1%) | .738 |
| Married | 34 (27.6%) | 18 (29%) | 16 (26.2%) | .731 |
| Divorced | 1 (0.8%) | 0 (0%) | 1 (1.6%) | .315 |
| Prefer Not to Say | 1 (0.8%) | 1 (1.6%) | 0 (0%) | .323 |
| Education | | | | |
| High School or Equivalent | 8 (6.5%) | 3 (4.8%) | 5 (8.2%) | .454 |
| Trade School | 1 (0.8%) | 1 (1.6%) | 0 (0%) | .323 |
| Some College | 19 (15.4%) | 9 (14.5%) | 10 (16.4%) | .776 |
| Associate Degree | 7 (5.7%) | 2 (3.2%) | 5 (8.2%) | .238 |
| Bachelor's Degree | 57 (46.3%) | 32 (51.6%) | 25 (41%) | .241 |
| Master's Degree | 28 (22.8%) | 15 (24.2%) | 13 (31.3%) | .706 |
| Doctoral Degree | 3 (2.4%) | 0 (0%) | 3 (4.9%) | .078 |
| BMI (median) | $27.8 \pm 10.8$ | $26.8 \pm 9.6$ | $29.9 \pm 11.8$ | .044* |
| Underweight (>18.5) | 3 (2.4%) | 2 (3.2%) | 1 (1.6%) | .572 |
| Normal weight (18.5-24.9) | 40 (32.5%) | 22 (35.5%) | 18 (29.5%) | .483 |
| Overweight (25-30) | 32 (26%) | 19 (29%) | 14 (23%) | .446 |
| <i>Obese (30+)</i> | 48 (39%) | 20 (32.3%) | 28 (45.9%) | .123 |
| Eating Disorder History^ | 18 (14.6%) | 9 (14.5%) | 9 (14.8%) | .974 |
| Anorexia Nervosa | 3 (2.4%) | 1 (1.6%) | 2 (3.3%) | .234 |
| Bulimia Nervosa | 4 (3.3%) | 2 (3.2%) | 2 (3.3%) | .974 |
| Binge Eating Disorder | 1 (0.8%) | 1 (1.6%) | 0 (0%) | .046* |
| Other Specified Feeding/Eating Disorder | 6 (4.9%) | 3 (4.8%) | 3 (4.9%) | .968 |
| Unspecified Feeding/Eating Disorder | 1 (0.8%) | 1 (1.6%) | 0 (0%) | .046* |
| Multiple | 3 (2.4%) | 1 (1.6%) | 2 (3.3%) | .234 |

<sup>\*</sup> Group difference at the 0.05 level ^ No participants had current eating disorders

Figure 1. CONSORT Flow Diagram



### References

- [1] Atalay, S., Baş, M., Eren, B., Karaca, E. and Baş, D. (2020). Intuitive eating, diet quality, body mass index and abnormal eating: A cross-sectional study in young Turkish women. *Progress in Nutrition*, 22(4). doi: 10.23751/pn.v22i4.9773
- <sup>[2]</sup>Bacon, L., & Aphramor, L. (2011). Weight science: Evaluating the evidence for a paradigm shift. *Nutrition Journal*, 10(9).
- [3] Barad, A., Cartledge, A., Gemmill, K., Misner, N. M., Santiago, C. E., Yavelow, M., & Langkamp-Henken, B. (2019). Associations between intuitive eating behaviors and fruit and vegetable intake among college students. *Journal of Nutrition Education and Behavior*, *51*(6), 758-762. doi: 10.1016/j.jneb.2019.03.010
- [4] Bombak, A., Monaghan, L. F., & Rich, E. (2018). Dietary approaches to weight-loss, health at every size, and beyond: Rethinking the war on obesity. *Social Theory and Health*, *17*, 89-108. doi: 10.1057/s41285-018-0070-9
- [5] Bond, F. W., Hayes, S. C., Baer, R. A., Carpenter, K. M., Guenole, N., Orcutt, H. K., Waltz, T., & Zettle, R. D. (2011). Preliminary psychometric properties of the Acceptance and Action Questionnaire II: A revised measure of psychological flexibility and experiential avoidance. *Behavior Therapy*, 42, 676-688.
- [6] Bruce, L. J., & Ricciardelli, L. A. (2016). A systematic review of the psychosocial correlates of intuitive eating among adult women. *Appetite*, *96*, 454-472. doi: 10.1016/j.appet.2015.10.012
- <sup>[7]</sup> Burnette, C. B., & Mazzeo, S. E. (2020). An uncontrolled pilot feasibility trial of an intuitive eating intervention for college women with disordered eating delivered through group and guided self-help modalities. *International Journal of Eating Disorders*, 1-13. doi: 10.1002/eat.23319
- [8] Byrne, S. M, Allen, K. L, Dove, E. R., Watt, F. J., & Nathan, P. R. (2008). The reliability of the dichotomous thinking in eating disorders scale. *Eating Behaviors*, *9*(2), 154-162. doi: 10.1016/j.eatbeh.2007.07.002
- <sup>[9]</sup> Clifford, D., Ozier, A., Bundros, J., Moore, J., Kreiser, A., & Morris, M. N. (2015). Impact of non-diet approaches on attitudes, behaviors, and health outcomes: A systematic review. *Journal of Nutrition Education and Behavior*, *47*, 143-155. doi: 10.1016/j.jneb.2014.12.002
- [10] Cole, R. E., & Horacek, T. (2010). Effectiveness of the "My Body Knows When" intuitive-eating pilot program. *American Journal of Health Behavior*, *34*(3), 286-297. doi:10.5993/ajhb.34.3.4.
- [11] Crow, S. J., Agras, W. S., Halmi, K., Mitchell, J. E., & Kraemer, H. C. (2002). Full syndromal versus subthreshold anorexia nervosa, bulimia nervosa, and binge eating disorder: A multicenter study. *International Journal of Eating Disorders*, 32(3), 309–318. doi: 10.1002/eat.10088
- [12] Deloitte Access Economics (2020). The social and economic cost of eating disorders in the United States of America: A report for the strategic training initiative for the prevention of eating disorders and the academy for eating disorders. Retrieved from: https://www.hsph.harvard.edu/striped/report-economic-costs-of-eating-disorders/.
- [13] Dwyer, J., Picciano, M. F., & Raiten, D. J. (2003). Collection of food and dietary supplement intake data: What we eat in America NHANES. *The Journal of Nutrition*, *133*(2), 590S-600S. doi: 10.1093/jn/133.2.590S
- [14] Hawks, S., Madanat, H., Hawks, J., & Harris, A. (2013). The relationship between intuitive eating and health indicators among college women. *Journal of Health Education*, *36*(6), 331-336, doi: 10.1080/19325037.2005.10608206
- [15] Hazzard, V. M., Telke, S. E., Simone, M., Anderson, L. M., Larson, N. I., & Neumark-Sztainer, D. (2020). Intuitive eating longitudinally predicts better psychological health and lower use of disordered eating behaviors: Findings from EAT 2010-2018. *Eating and Weight Disorders*. doi: 10.1007/s40519-020-00852-4

- [16] Horwath, C., Hagmann, D., & Hartmann, C. (2019). Intuitive eating and food intake in men and women: Results from the Swiss food panel study. *Appetite*, *135*, 61-71. doi: 10.1016/j.appet.2018.12.036
- [17] Finkelstein, E. A., Trogdon, J. G., Cohen, J. W., & Dietz, W. (2009). Annual medical spending attributable to obesity: Payer and service specific estimates. *Health Affairs*, 28(5), 822-831. doi: 10.1377/hlthaff.28.5.w822
- [18] Fitzsimmons-Craft, E. E. (2011). Social psychological theories of disordered eating in college women: Review and integration. *Clinical Psychology Review*, *31*(7), 1224–1237. doi: 10.1016/j.cpr.2011.07.011
- [19] Galmiche, M., Dechelotte, P., Lambert, G., & Tavolacci, M. P. (2019). Prevalence of eating disorders over the 2000-2018 period: A systematic literature review. *American Journal of Clinical Nutrition*, 109, 1402-1413. doi: 10.1093/ajcn/nqy342.
- <sup>[20]</sup> Hales, C. M., Carroll, M. D., Fryar, C. D., & Ogden, C. L. (2020). Prevalence of obesity and severe obesity among adults: United States, 2017-2018. *National Center for Health Statistics Data Brief*, *360*. U.S. Department of Health and Human Services.
- [21] Howard, B. V., Manson, J. E., Beresford, S. A., Frank, G., Jones, B., Rodabough, R. J., Snetselaar, L., Thomson, C., Tinker, L., Vitolins, M., & Prentice, R. (2006). Low-fat dietary pattern and weight change over 7 years: The women's health initiative dietary modification trial. *The Journal of American Medical Association*, 295(1), 39-49. doi: 10.1001/jama.295.1.39
- [22] Kerin, J. L., Webb, H. J., & Zimmer-Gembeck, M. J. (2019). Intuitive, mindful, emotional, external and regulatory eating behaviours and beliefs: An investigation of the core components. *Appetite*, *132*, 139-146. doi: 10.1016/j.appet.2018.10.011
- <sup>[23]</sup> Lauzon, B. D., Romon, M., Deschamps, V., Lafay, L., Borys, J. M., Karlsson, J., Ducimetere, P., & Charles, M. A. (2004). The three-factor eating questionnaire-r18 is able to distinguish among different eating patterns in a general population. *Nutritional Epidemiology*, 2372-2380.
- [24] Linardon, J., & Mitchell, S. (2017). Rigid dietary control, flexible dietary control, and intuitive eating: Evidence for their differential relationship to disordered eating and body image concerns. *Eating Behaviors*, 26, 16-22. doi: 10.1016/j.eatbeh.2017.01.008
- <sup>[25]</sup>Lipson, S. K., Jones, J. M., Taylor, C. B., Wilfley, D. E., Eichen, D. M., Fitzsimmons-Craft, E. E., & Eisenberg, D. (2017). Understanding and promoting treatment-seeking for eating disorders and body image concerns on college campuses through online screening, prevention and intervention. *Eating Behaviors*, *25*, 68–73. doi: 10.1016/j.eatbeh.2016.03.020
- [26] Madden, C. E., Leong, S. L., Gray, A., & Horwath, C. C. (2012). Eating in response to hunger and satiety signals is related to BMI in a nationwide sample of 1601 mid-age New Zealand women. *Public Health Nutrition*, *15*(12), 2272–2279 doi:10.1017/S1368980012000882
- [27] Martin, C. B., Herrick, K. A., Sarafrazi, N., & Ogden, C. L. (2018). Attempts to lose weight among adults in the United States, 2013-2016. *National Center for Health Statistics Data Brief*, 313. U.S. Department of Health and Human Services.
- <sup>[28]</sup>Neumark-Sztainer, D. R., Wall, M., Larson, N. I., Eisenberg, M. E., & Loth, K. (2011). Dieting and disordered eating behaviors from adolescence to young adulthood: Findings from a 10-year longitudinal study. *Journal of the American Dietetic Association*, 111(7), 1004–1011. doi: 10.1016/j.jada.2011.04.012
- [29] O'Hara, L., & Gregg, J. (2012). Human rights casualties from the "war on obesity": Why focusing on body weight is inconsistent with a human rights approach to health. *Fat Studies*, *1*, 32-46. doi: 10.1080/21604851.2012.627790
- [30] Pereira, R. F., & Alvarenga, M. (2007). Disordered eating: Identifying, treating, preventing, and differentiating it from eating disorders. *Diabetes Spectrum*, 20(3), 141-148.
- [31] Reba-Harrelson, L., Von Holle, A., Hamer, R. M., Swann, R., Reyes, M. L., & Bulik, C. M. (2009). Patterns and prevalence of disordered eating and weight control behaviors in women ages 25-45. *Eating and Weight Disorders*, *14*(4), 190-198.

- [32] Ruzanska, U. A., & Warschburger, P. (2020). How is intuitive eating related to self-reported and laboratory food intake in middle-aged adults?. *Eating Behaviors*, *38*. doi: 10.1016/j.eatbeh.2020.101405
- [33] Salas, X. R. (2015). The ineffectiveness and unintended consequences of the public health war on obesity. *Canadian Journal of Public Health*, 106(2), 79-81. doi: 10.17269/CJPH.106.4757
- [34] Schaefer, J. T., & Magnuson, A. B. (2014). A review of interventions that promote eating by internal cues. *Academy of Nutrition and Dietetics*, 114(5), doi: 10.1016/j.jand.2013.12.024
- [35] Tribole, E., & Resch, E. (2003). *Intuitive eating: A revolutionary program that works*. St. Martin's Griffin: New York, New York.
- [36] Tylka, T. L., Calogero, R. M., & Danielsdóttir, S. (2020). Intuitive eating is connected to self-reported weight stability in community women and men. *Eating Disorders*, 28(3), 256-264. doi: 10.1080/10640266.2019.1580126
- [37] Tylka, T. L., & Van Diest, A. M. (2013). The Intuitive Eating Scale-2: Item refinement and psychometric evaluation with college women and men. *Journal of Counseling Psychology*, 60(1), 137-153. doi: 10.1037/a0030893
- [38] Tylka & Wood-Barcalow, N. L. (2015). The body appreciation scale-2: Item refinement and psychometric evaluation. *Body Image*, *12*, 53-67. doi: 10.1016/j.bodyim.2014.09.006
- [39] Van Dyke, N., & Drinkwater, E. J. (2013). Relationships between intuitive eating and health indicators: Literature review. *Public Health Nutrition*, *17*(8), 1757-66. doi: 10.1017/S1368980013002139
- <sup>[40]</sup> Wilson, R. E., Marshall, R. D., Murkami, J. M, & Latner, J. D. (2020). Brief non-dieting intervention increases intuitive eating and reduces dieting intention, body image dissatisfaction, and anti-fat attitudes: A randomized controlled trial. *Appetite*, *148*(1). doi: 10.1016/j.appet.2019.104556
- [41] White, S., Reynolds-Malear, J. B., & Cordero, E. (2011). Disordered eating and the use of unhealthy weight control methods in college students: 1995, 2002, and 2008. *Eating Disorders*, 19(4), 323-334. doi: 10.1080/10640266.2011.584805